CLINICAL TRIAL: NCT03338894
Title: A Controlled Trial of Yoga in Pediatric Inflammatory Bowel Disease (IBD)
Brief Title: A Trial of Yoga in Pediatric Inflammatory Bowel Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Atlantic Health System (Other)
Responsible Party: Principal Investigator, Alycia Leiby, MD, Principal Investigator, Atlantic Health System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: YOGAL
Record Dates: First submitted 2017-11-07; First posted 2017-11-09 (Actual); Results first posted 2021-06-08 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Inflammatory Bowel Disease; Crohn's Disease; Ulcerative Colitis
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative | interventions — Yoga

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Yoga group (Other): Each subject will serve as their own control
  Interventions: Behavioral: Yoga

INTERVENTIONS:
Behavioral: Yoga — 1 Hour yoga class

SUMMARY:
IBD adds additional stressors as a chronic disease that has unpredictable and sometimes embarrassing symptoms to the normal challenges that teenagers face. Stress and how stressful events are perceived, may contribute to worsening of disease. Complementary and alternative medicine (CAM), are used often by pediatric IBD patients and maybe beneficial in decreasing stress and improving quality of life. Yoga could be a well suited paring with standard medical therapy to decrease and provide a better sense of control and improve quality of life.

DETAILED DESCRIPTION:
Approximately 25% of Inflammatory bowel disease (IBD) is diagnosed in the pediatric age group, with the peak age of onset in the adolescent years. IBD adds additional stressors of a chronic disease with unpredictable and potentially embarrassing symptoms to the expected challenges of psychological and social adjustment that teenagers face. Various techniques, such as psychotherapy programs and IBD overnight camp experiences, have been studied to decrease psychological distress and improve quality of life. Stress, and particularly how stressful events are perceived, may play a role in triggering IBD flares. Complementary and alternative medicine (CAM), especially mind-body techniques are used often by pediatric IBD patients and may be beneficial in decreasing stress and improving quality of life (QOL). Yoga may be well suited as an adjunct to conventional IBD therapy to decrease stress, provide a greater sense of bodily control and improve QOL.

The primary goal of this project is to determine if a structured Yoga program, in addition to standard medical therapy, improves HRQOL in pediatric patients diagnosed with inflammatory bowel disease (IBD). Investigators will also examine if the yoga program improves self efficacy, which is a person's belief about their ability to influence events that affect their lives. Disease response and remission rates will be followed as well, in order to stratify HRQOL outcomes in the yoga group.

Patients will each serve as their own control and complete questionnaires at enrollment and at the start and end of the 12 week group yoga class sessions. They will also complete the questionnaires three months after finishing the class sessions. .The program will consist of a live group class session over 12 weeks. Baseline and follow-up questionnaires will be used to determine there are changes in QOL, self-efficacy, and disease response.

ELIGIBILITY:
Inclusion Criteria:

* Both males and females patients with IBD
* Ages 10-17 years
* Not currently practicing specific mind-body techniques (yoga, pranayama - deep breathing, biofeedback, hypnosis, guide imagery)
* Diagnosis of IBD

Exclusion Criteria:

* Other chronic systemic disease ex. Rheumatoid arthritis, Cystic fibrosis, Celiac or chronic neurologic conditions

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 78 (Actual)
Dates: Start 2017-12-13 (Actual); Primary Completion 2020-03-18 (Actual); Study Completion 2021-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alycia Leiby, MD, Principal Investigator — Atlantic Health/Goryeb Children's Hospital
Locations (2):
- United States (2):
  - Morristown Memorial Hospital/Goyerb Children's Hospital, Morristown, New Jersey
  - Children's Hospital of Philadelphia/Roberts Center for Pediatric Research, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shepanski MA, Hurd LB, Culton K, Markowitz JE, Mamula P, Baldassano RN. Health-related quality of life improves in children and adolescents with inflammatory bowel disease after attending a camp sponsored by the Crohn's and Colitis Foundation of America. Inflamm Bowel Dis. 2005 Feb;11(2):164-70. doi: 10.1097/00054725-200502000-00010. PMID 15677910
- [Background] McCormick M, Reed-Knight B, Lewis JD, Gold BD, Blount RL. Coping skills for reducing pain and somatic symptoms in adolescents with IBD. Inflamm Bowel Dis. 2010 Dec;16(12):2148-57. doi: 10.1002/ibd.21302. PMID 20848505
- [Background] Singh S, Graff LA, Bernstein CN. Do NSAIDs, antibiotics, infections, or stress trigger flares in IBD? Am J Gastroenterol. 2009 May;104(5):1298-313; quiz 1314. doi: 10.1038/ajg.2009.15. Epub 2009 Mar 31. PMID 19337242
- [Background] Wong AP, Clark AL, Garnett EA, Acree M, Cohen SA, Ferry GD, Heyman MB. Use of complementary medicine in pediatric patients with inflammatory bowel disease: results from a multicenter survey. J Pediatr Gastroenterol Nutr. 2009 Jan;48(1):55-60. doi: 10.1097/MPG.0b013e318169330f. PMID 19172124
- [Background] Markowitz JE, Mamula P, delRosario JF, Baldassano RN, Lewis JD, Jawad AF, Culton K, Strom BL. Patterns of complementary and alternative medicine use in a population of pediatric patients with inflammatory bowel disease. Inflamm Bowel Dis. 2004 Sep;10(5):599-605. doi: 10.1097/00054725-200409000-00015. PMID 15472521
- [Background] Heuschkel R, Afzal N, Wuerth A, Zurakowski D, Leichtner A, Kemper K, Tolia V, Bousvaros A. Complementary medicine use in children and young adults with inflammatory bowel disease. Am J Gastroenterol. 2002 Feb;97(2):382-8. doi: 10.1111/j.1572-0241.2002.05474.x. PMID 11866277
- [Background] Day AS, Whitten KE, Bohane TD. Use of complementary and alternative medicines by children and adolescents with inflammatory bowel disease. J Paediatr Child Health. 2004 Dec;40(12):681-4. doi: 10.1111/j.1440-1754.2004.00510.x. PMID 15569284
- [Background] Cotton S, Humenay Roberts Y, Tsevat J, Britto MT, Succop P, McGrady ME, Yi MS. Mind-body complementary alternative medicine use and quality of life in adolescents with inflammatory bowel disease. Inflamm Bowel Dis. 2010 Mar;16(3):501-6. doi: 10.1002/ibd.21045. PMID 19705417
- [Background] Kuttner L, Chambers CT, Hardial J, Israel DM, Jacobson K, Evans K. A randomized trial of yoga for adolescents with irritable bowel syndrome. Pain Res Manag. 2006 Winter;11(4):217-23. doi: 10.1155/2006/731628. PMID 17149454
- [Background] Otley A, Smith C, Nicholas D, Munk M, Avolio J, Sherman PM, Griffiths AM. The IMPACT questionnaire: a valid measure of health-related quality of life in pediatric inflammatory bowel disease. J Pediatr Gastroenterol Nutr. 2002 Oct;35(4):557-63. doi: 10.1097/00005176-200210000-00018. PMID 12394384
- [Background] Hyams J, Markowitz J, Otley A, Rosh J, Mack D, Bousvaros A, Kugathasan S, Pfefferkorn M, Tolia V, Evans J, Treem W, Wyllie R, Rothbaum R, del Rosario J, Katz A, Mezoff A, Oliva-Hemker M, Lerer T, Griffiths A; Pediatric Inflammatory Bowel Disease Collaborative Research Group. Evaluation of the pediatric crohn disease activity index: a prospective multicenter experience. J Pediatr Gastroenterol Nutr. 2005 Oct;41(4):416-21. doi: 10.1097/01.mpg.0000183350.46795.42. PMID 16205508
- [Background] Hyams J, Markowitz J, Lerer T, Griffiths A, Mack D, Bousvaros A, Otley A, Evans J, Pfefferkorn M, Rosh J, Rothbaum R, Kugathasan S, Mezoff A, Wyllie R, Tolia V, delRosario JF, Moyer MS, Oliva-Hemker M, Leleiko N; Pediatric Inflammatory Bowel Disease Collaborative Research Group. The natural history of corticosteroid therapy for ulcerative colitis in children. Clin Gastroenterol Hepatol. 2006 Sep;4(9):1118-23. doi: 10.1016/j.cgh.2006.04.008. Epub 2006 Jul 3. PMID 16820327
- [Background] Markowitz J, Hyams J, Mack D, Leleiko N, Evans J, Kugathasan S, Pfefferkorn M, Mezoff A, Rosh J, Tolia V, Otley A, Griffiths A, Moyer MS, Oliva-Hemker M, Wyllie R, Rothbaum R, Bousvaros A, Del Rosario JF, Hale S, Lerer T; Pediatric IBD Collaborative Research Group. Corticosteroid therapy in the age of infliximab: acute and 1-year outcomes in newly diagnosed children with Crohn's disease. Clin Gastroenterol Hepatol. 2006 Sep;4(9):1124-9. doi: 10.1016/j.cgh.2006.05.011. Epub 2006 Jul 24. PMID 16861053

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study enrollment was offered during office or infusion visit. Recruitment began December 2017 and closed August 2019.
Period: Overall Study
Arm/Group | Yoga Group
Started | 78
Completed | 56
Not Completed | 22
Not completed — Withdrew, or not able to attend 9 or more classes, or did not complete final survey. | 22

BASELINE CHARACTERISTICS:
Arm/Group | Yoga Group
Number analyzed (Participants) | 56
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 13 [12 to 15]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39
  Male | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 49
  Unknown or Not Reported | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 42
  More than one race | 0
  Unknown or Not Reported | 10
Region of Enrollment [Number; unit: participants]
  United States | 56
Inflammatory Bowel Disease Type [Count of Participants; unit: Participants]
  Crohn's Disease | 41
  Ulcerative Colitis/Inflammatory Bowel Disease unspecified | 15

OUTCOME MEASURES:

1. Primary Outcome: Pediatric Quality of Life Inventory
Description: The number of patients diagnosed with Inflammatory Bowel disease that have shown an improved health related quality of life (HRQOL) as assessed by the Pediatric Quality of Life survey after a structured yoga program, comparing pre-yoga HRQOL to post-yoga HRQOL. The Peds QOL age related surveys are validated pediatric questionnaires that measure general HRQOL in children ages 8-17 years. They consist of 23 questions in areas of social, school, emotional and physical functioning. The answers are scored on a 5 point scale and then reverse scored and linearly transformed to a scale of 1-100 scale.
Time Frame: Compared difference from enrollment (time0) to start yoga class (time1), to difference from first yoga class (time1) to last yoga class (time2) 90 days, difference from first yoga class (time1) to 3 months after last yoga class (time 3) 180 days.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Yoga Group
Number analyzed (Participants) | 54
score on a scale
  time 0 to time 1 | 2.14 (8.79)
  time 1 to time 2 | 1.5 (8.01)
  time 1 to time 3 | 2.8 (10.24)

2. Secondary Outcome: General Perceived Self Efficacy Scale
Description: This is a 10 item scale that measures a patient's general sense of perceived self-efficacy, aiming to predict coping with daily life as well as adaptation after stressful life events. The General Self Efficacy Scale is correlated to emotion, optimism, and work satisfaction. Negative coefficients were found for depression, stress, health complaints, burnout and anxiety. The total score is calculated by finding the sum of all item. For the General Self-Efficacy, the total score ranges between 10 to 40, with a higher score indicating more self-efficacy.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Yoga Group
Number analyzed (Participants) | 54
score on a scale
  Time 0 to Time 1 | 0.27 (3.89)
  Time 1 to Time 2 | 0.4 (4.32)
  Time 1 to Time 3 | 1 (3.603)

ADVERSE EVENTS:
Time Frame: 6 month
Arm/Group | Yoga Group
All-Cause Mortality (participants affected / at risk) | 0/56
Serious Adverse Events (participants affected / at risk) | 0/56
Other Adverse Events (participants affected / at risk) | 0/56

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-14): https://cdn.clinicaltrials.gov/large-docs/94/NCT03338894/Prot_SAP_000.pdf